CLINICAL TRIAL: NCT03501121
Title: Extended Follow up of the TARGIT-A Trial
Acronym: TARGIT-X
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0774
Record Dates: First submitted 2018-03-15; First posted 2018-04-18 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Breast Neoplasm Female
Keywords: intra-operative radiation therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All UK patients who participated in the TARGIT-A Trial were initially treated for early breast cancer between 2000-2012. A total of 3451 patients from 33 hospitals in 11 countries participated in the trial and a comparison was made between traditional radiotherapy given over several weeks (external beam radiotherapy, EBRT) with TARGeted Intraoperative radioTherapy (TARGIT-IORT) as a single dose given during the operation to remove the breast cancer. The trial was funded by the Health Technology Assessment (HTA) programme of the Department of Health, UK and sponsored by University College London. The results from this trial have been published in major medical journals and have already started changing the way breast cancer in treated around the world; please see www.targit.org.uk for more details. We would like to continue to collect data about the health status of all patients to enable us to learn about longer term differences in the effects of these treatments on health. An analysis of this information could improve treatment for patients with breast cancer. For this, HTA have granted us further funding.

ELIGIBILITY:
Inclusion Criteria:

* All patients who participated in the TARGIT-A trial (NCT00983684).

Exclusion Criteria:

* Any patient who has withdrawn consent for further follow-up, or died.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who participated in the TARGIT-A trial (see NCT00983684).
Sampling Method: Non-Probability Sample
Enrollment: 714 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Long-term follow-up through direct patient contact | 60 months
  Maintaining regular contact with subjects to obtain self-reported health status in order to collect long-term follow-up of patients participating in the TARGIT A Trial.

SECONDARY OUTCOMES:
Long-term follow-up through national registries | Up to 20 years
  Collect death & new primary cancer data from UK patients through the Office for National Statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Vaidya, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - University College London, London
  - Royal Hampshire County Hospital, Winchester